CLINICAL TRIAL: NCT01370629
Title: A Prospective Observational Registry Study to Characterise Normal Conditions of Use, Dosing and Safety Following Administration of Vernakalant IV Sterile Concentrate
Brief Title: Study of Normal Conditions of Use, Dosing, and Safety of Intravenous (IV) Administration of Vernakalant (MK-6621-049)
Status: Completed | Type: Observational
Sponsor: Correvio International Sarl (Industry)
Responsible Party: Sponsor
Organization: Advanz Pharma (Industry)
Other Study IDs: 6621-049; EP01029.004 (Other: Merck)
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All participants: Participants treated with vernakalant IV in acute care and inpatient hospital settings
  Interventions: Drug: Vernakalant

INTERVENTIONS:
Drug: Vernakalant — Prescribed at the discretion of the physician in accordance with their usual practice
  Other Names: BRINAVESS®

SUMMARY:
This non-interventional prospective study is a post-authorization safety study (PASS) of vernakalant conducted to collect information about normal conditions of use and appropriate dosing, and to quantify possible medically significant risks associated with the use of vernakalant in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* To be treated with intravenous vernakalant, independently of this study
* Participant and/or legal guardians willing to provide informed consent and/or informed assent according to local regulations

Exclusion Criteria:

- Enrollment in an investigational drug or device clinical trial in the 30 days prior to study enrolment. Participation in another non-interventional drug or device study or registry is permitted.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants treated with intravenous vernakalant in acute care and inpatient hospital settings per usual care
Sampling Method: Non-Probability Sample
Enrollment: 2015 (Actual)
Dates: Start 2011-08; Primary Completion 2018-04-05 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Medizinische Universitat Wien, Vienna, Austria
- Aalborg, Denmark
- Kuopio Hospital, Kuopio, Finland
- St-Vincenz Krankenhaus, Paderborn, Germany
- Hospital Universitario Severo Ochoa, Madrid, Spain
- Skanes Universistetssjukhus, Malmo, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 2015
Completed | 2009
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 2009
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1024
  >=65 years | 985
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 787
  Male | 1222
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 1931
  Race: Black | 5
  Race: Hispanic | 6
  Race: Asian | 2
  Race: Other | 65
Region of Enrollment [Number; unit: participants]
  Austria | 547
  Sweden | 493
  Finland | 256
  Denmark | 113
  Germany | 300
  Spain | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Significant Hypotension
Description: Significant hypotension is defined as: symptomatic hypotension with systolic blood pressure (BP) <90 mmHg, requiring treatment with vasopressors
Time Frame: Start (baseline) of first vernakalant infusion up to 24 hours after the last infusion
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 2009
Participants | 2

2. Primary Outcome: Number of Participants Experiencing Significant Ventricular Arrhythmia
Time Frame: Start (baseline) of first vernakalant infusion up to 24 hours after the last infusion
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 2009
Participants | 1

3. Primary Outcome: Number of Participants Experiencing Significant Atrial Flutter
Time Frame: Start (baseline) of first vernakalant infusion up to 24 hours after the last infusion
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 2009
Participants | 2

4. Primary Outcome: Number of Participants Experiencing Significant Bradycardia
Time Frame: Start (baseline) of first vernakalant infusion up to 24 hours after the last infusion
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 2009
Participants | 15

5. Secondary Outcome: Number of Participants Who Are Converted to Sinus Rhythm for at Least One Minute
Time Frame: Up to 90 minutes after the start (baseline) of first infusion of vernakalant
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 1936
Participants | 1359

ADVERSE EVENTS:
Time Frame: 24 hours after the last infusion of vernakalant IV or until discharge / end of medical encounter, whichever occurred earlier
Description: Health outcomes of interest (HOIs) were reported as defined in the study protocol section
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/2009
Serious Adverse Events (participants affected / at risk) | 26/2009
Other Adverse Events (participants affected / at risk) | 62/2009
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=2009)
Significant hypotension (Cardiac disorders) | 2 (2) — Significant hypotension defined as: symptomatic hypotension with systolic blood pressure (BP) <90 mmHg, requiring treatment with vasopressors
significant ventricular arrhythmia (Cardiac disorders) | 1 (1) — Significant ventricular arrhythmia: Sustained VT with a ventricular heart rate >120 bpm >30 seconds or VT that required intervention or Torsade de Pointes with a duration of >10 seconds, or Ventricular fibrillation of any duration
Significant bradycardia (Cardiac disorders) | 15 (15) — Significant bradycardia defined as: bradycardia requiring electrical pacing (temporary or permanent) or any other serious adverse event (SAE) reports involving bradycardia
Significant atrial flutter with 1:1 conduction (Cardiac disorders) | 1 (1) — Significant atrial flutter (AFL) defined as: AFL with 1:1 atrioventricular conduction of >10 seconds duration and a ventricular rate of >200 bpm
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1)
Non-sustained wide QRS complex tachycardia (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=2009)
Dysgeusia (Nervous system disorders) | 35 (35)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT01370629/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT01370629/SAP_001.pdf